CLINICAL TRIAL: NCT06558448
Title: Developing a Prognostic Warning System for Heart Failure Based on Multimodal Clinical Data: a Multi-center Retrospective Study
Brief Title: Multimodal Prognostic System for Heart Failure: A Multi-Center Study
Status: Not yet recruiting | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, QianQian Wang, student, Chongqing Medical University
Other Study IDs: CYS240347
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter retrospective research aimed at developing a heart failure prognosis warning system based on multimodal clinical data to improve the diagnosis and treatment of heart failure.

This study aims to address the following main questions:

1. What are the clinical characteristics and current treatment status of heart failure patients?
2. What factors influence the onset of heart failure and the prognosis of patients?
3. How can real-world big data be utilized to construct an accurate heart failure prognosis assessment model?
4. How can this prognosis assessment model help improve the therapeutic effects and quality of life for heart failure patients?

ELIGIBILITY:
Inclusion Criteria:

Age Requirement: We plan to include adult patients aged 18 and above to ensure the study covers a broad spectrum of the adult heart failure patient population.

Diagnostic Criteria: Patients should have a discharge diagnosis of heart failure according to the guidelines for heart failure diagnosis and treatment.

Time Frame: The discharge time of patients should be between January 2011 and December 2024 to collect and analyze data from the past several years.

Data Integrity: There is a preference for including medical records with high data integrity, but the specific criteria may be adjusted according to the actual situation of the dataset.

Exclusion Criteria:

Data Missing: Patients with more than 30% missing data in their medical records may be considered for exclusion to ensure the accuracy and reliability of the analysis.

Diagnostic Inconsistency: Patients with unclear diagnoses or potential for confusion with other diseases may be excluded to ensure the specificity of the study.

Non-standard Treatment: Patients who have not received treatment according to the established treatment protocol may be excluded to reduce the impact of treatment variability on the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this research consists of adult patients, aged 18 and above, with a discharge diagnosis of heart failure between January 2011 and December 2024, as per the guidelines for the diagnosis and treatment of heart failure . The patients' electronic medical records, which include demographic information, comorbidities, treatment plans, and various clinical indicators, are sourced , ensuring a comprehensive and in-depth analysis of the heart failure patient cohort.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality or other adverse outcomes, including readmission, in-hospital infection, respiratory failure, liver failure, and renal failure. | Evaluations will be conducted within 30, 60, or 90 days post-admission for heart failure patients to assess the impact of the condition and the effectiveness of treatment.
  The study focuses on evaluating the risk factors and predictors of in-hospital mortality and various adverse outcomes in heart failure patients, encompassing events such as readmission due to exacerbation of the condition, infections acquired during hospital stay, critical impairments in respiratory, liver, and kidney functions that may complicate the clinical course and impact patient prognosis.

IPD SHARING:
Plan to Share IPD: No
The data analyzed in this study are subject to the following licenses/restrictions: due to ethics committee regulations, the access to the dataset supporting the findings of this study is limited and not public. Requests to access these datasets should be directed to XZ Liu(xiaozhuliu2021@163.com).